CLINICAL TRIAL: NCT06355908
Title: Safety, Tolerability and Efficacy of Enhanced IL-13Rα2 Targeted Chimeric Antigen Receptor T Cell Immunotherapy Against Recurrent/Refractory Grade 4 Glioma
Brief Title: IL13Rα2 CAR-T for Patients With r/r Glioma
Acronym: ENHANCING
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Temporarily suspended for HGRAC filing requirements
Sponsor: Yang Zhang (Other)
Collaborators: TCRCure Biopharma Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Yang Zhang, Clinical Professor, Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TT002
Record Dates: First submitted 2024-03-23; First posted 2024-04-10 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Glioma
Keywords: r/r WHO4 glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IL13Rα2 CAR-T (Experimental): Biological: IL13Rα2 CAR-T
  Interventions: Biological: IL13Rα2 CAR-T

INTERVENTIONS:
Biological: IL13Rα2 CAR-T — The IL13Rα2 CAR-T cells will be administered via intraventricular infusion every 2 weekly via an Ommaya reservoir.

SUMMARY:
This is a dose exploration clinical trial to assess the safety and feasibility of the IL13Ra2-targeted CAR-T in glioma.

DETAILED DESCRIPTION:
Interleukin 13 receptor subunit alpha-2 (IL13Ra2A) is a high-affinity membrane receptor of the anti-inflammatory Th2 cytokine IL13, which is overexpressed in glioma and correlated with poor prognosis.

Chimeric antigen receptor (CAR) T cell therapy is a promising treatment approach for many malignancies. IL13Ra2-targeted CAR-T cells are under investigation in several clinical trials in primary CNS malignancies.

The investigators now designed a new structure CAR targeted IL13Ra2, and initiated a single arm, open, dose exploration clinical trial to evaluate the safety, tolerability, clinical efficacy, and pharmacokinetic characteristics of IL13Rα2 CAR-T for patients with glioma. This clinical trial will enroll 12-30 cases of patients with IL13α2-positive recurrent or refractory WHO grade 4 glioma (r/r WHO4 glioma), aiming to find the maximum tolerable dose (MTD), the recommended phase 2 dose (RP2D) and preliminary efficacy of the new structure IL13Ra2 CAR-T.

ELIGIBILITY:
Inclusion criteria:

1. Male or female aged 18-75 years (including 18 and 75 years old).
2. Karnofsky scale score (KPS)≥50.
3. Subjects with WHO grade 4 gliomas who have relapsed or progressed during or after standard treatments such as surgery, radiotherapy, and chemotherapy.
4. Tumor with IL13Rα2 positive expression.
5. Availability in collecting peripheral blood mononuclear cells (PBMCs).
6. Adequate laboratory values and adequate organ function.
7. Patients with childbearing/fathering potential must agree to use highly effective contraception.

Exclusion criteria:

1. Pregnant or breastfeeding females.
2. Contraindication to bevacizumab.
3. Within 5 days prior to the infusion of CAR-T cells, subjects receiving systemic administration of steroids with dosage more than 10mg/d prednisone or the equivalent doses of other steroids (not including inhaled corticosteroid).
4. Comorbid with other uncontrolled malignancy.
5. Active immunodeficiency virus (HIV) or hepatitis B virus or hepatitis C virus or tuberculosis infection.
6. Autoimmune diseases.
7. Severe or uncontrolled psychiatric diseases or condition that could increase adverse events or interfere the evaluation of outcomes.
8. Subjects who have previously received cell therapy (such as TCR-T, CAR-T, TIL, etc.).
9. Subjects with other conditions that would interfere trial participation at the investigator's discretion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Safety of IL13Rα2 CAR-T | Day 0 - Day 730
  The safety of IL13Rα2 CAR-T will be assessed based on the totality of dose-limiting toxicity (DLT) and adverse event (AE) data collected during this phase.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Day 0 - Day 730
  To evaluate the percentage of subjects who have a confirmed partial response (PR) and complete response (CR) per immunotherapy response assessment in neuro-oncology (iRANO) criteria.
Duration of Response (DOR) | Day 0 - Day 730
  To evaluate the duration from the time that criteria are met for CR or PR per iRANO until disease progression or death due to any cause.
Progression Free Survival (PFS) | Day 0 - Day 730
  To evaluate the time from the date of the first CAR-T infusion until disease progression per iRANO or death due to any cause.
Overall Survival (OS) | Day 0 - Day 730
  To evaluate the time from the date of the first CAR-T infusion to death due to any cause.
Overall Survival (OS) at 6 months (OS6) | Day 0 - Day 180
  To evaluate the percentage of survival subjects at 6 months after the first CAR-T infusion.
Overall Survival (OS) at 12 months (OS12) | Day 0 - Day 365
  To evaluate the percentage of survival subjects at 12 months after the first CAR-T infusion.
The levels of IL13Rα2 CAR-T cell and IL13Rα2 CAR in the CSF and peripheral blood | Day 0 - Day 730
  To detect the levels of IL13Rα2 CAR-T cell and IL13Rα2 CAR in the CSF and peripheral blood.
The levels of cytokines in the CSF and peripheral blood | Day 0 - Day 730
  To detect levels of cytokines in the CSF and peripheral blood, cytokines will include IL-2, IL-6, IFN-γ, TNF-α, etc.

OTHER OUTCOMES:
The Exploratory Indicators | Day 0 - Day 730
  To analyze tumor microenvironment and CAR-T cell infiltrative levels in tumor tissues before and after treatment by immunohistochemistry and/or transcriptome sequencing, and explore the tumor or immune cell markers related to disease prognosis and IL13Rα2 expression.

CONTACTS AND LOCATIONS:
Overall Officials: Nan Ji, MD, PhD, Principal Investigator — Beijing Tiantan Hospital; Yang Zhang, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No